CLINICAL TRIAL: NCT00871286
Title: Role of Point-of-Care CT Scanning in Patients Presenting With Symptoms of Chronic Rhinosinusitis
Brief Title: Point-of-Care Computed Tomography (CT) Chronic Rhinosinusitis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rakesh Chandra, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 8997; STU 8997
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic rhinosinusitis; Chronic sinusitis; CRS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT scan (sinus) pre-tx (Experimental): Sinus CT scan performed at initial otolaryngology (ear, nose, and throat)visit
  Interventions: Procedure: Pre-treatment Sinus CT Scan
- CT scan (sinus) post-tx (Other): Sinus CT scan performed after 3-4 weeks of antibiotic treatment and any other indicated medical treatment(s), per insurance company guidelines
  Interventions: Procedure: Post-treatment Sinus CT Scan

INTERVENTIONS:
Procedure: Pre-treatment Sinus CT Scan — Pre-treatment Sinus CT Scan
  Arms: CT scan (sinus) pre-tx
Procedure: Post-treatment Sinus CT Scan — Post-treatment Sinus CT Scan
  Arms: CT scan (sinus) post-tx

SUMMARY:
The purpose of this research study is to determine whether or not computed tomography (CT) scans performed on patients with symptoms of chronic rhinosinusitis (CRS) but without any physical signs of the disease will (1) prove to be less expensive in the treatment and evaluation as compared to current practices, (2) avoid the use of unnecessary antibiotic prescriptions, and (3) provide a more efficient way to diagnose conditions in patients who have had CRS ruled out as a cause.

The investigators hypothesize that current guidelines, when applied to subjects with symptoms of CRS in the absence of physical signs may be associated with (1) increased unnecessary prescription of antibiotics, (2) delay in further essential workup, and (3) increased overall health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects actively meeting the symptomatic criteria for CRS as defined by the Taskforce on Rhinosinusitis but with physical and endoscopic examination that is within normal limits

Exclusion Criteria:

* Subjects who are pregnant
* Subjects with a diagnosis of immune suppression or suspicion of malignancy that may be affecting the nose/paranasal sinuses
* Subjects who have had prior sinus surgery or who have been previously treated with a >3 week course of broad spectrum antibiotics for CRS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh K Chandra, MD, Principal Investigator — Northwestern University, Northwestern Medical Faculty Foundation, Northwestern Memorial Hospital
Locations (1):
- Northwestern University/Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

REFERENCES:
- [Background] Stankiewicz JA, Chow JM. A diagnostic dilemma for chronic rhinosinusitis: definition accuracy and validity. Am J Rhinol. 2002 Jul-Aug;16(4):199-202. PMID 12222944
- [Background] Stankiewicz JA, Chow JM. Cost analysis in the diagnosis of chronic rhinosinusitis. Am J Rhinol. 2003 May-Jun;17(3):139-42. PMID 12862401
- [Background] Meltzer EO, Hamilos DL, Hadley JA, Lanza DC, Marple BF, Nicklas RA, Bachert C, Baraniuk J, Baroody FM, Benninger MS, Brook I, Chowdhury BA, Druce HM, Durham S, Ferguson B, Gwaltney JM Jr, Kaliner M, Kennedy DW, Lund V, Naclerio R, Pawankar R, Piccirillo JF, Rohane P, Simon R, Slavin RG, Togias A, Wald ER, Zinreich SJ; American Academy of Allergy, Asthma and Immunology; American Academy of Otolaryngic Allergy; American Academy of Otolaryngology-Head and Neck Surgery; American College of Allergy, Asthma and Immunology; American Rhinologic Society. Rhinosinusitis: Establishing definitions for clinical research and patient care. Otolaryngol Head Neck Surg. 2004 Dec;131(6 Suppl):S1-62. doi: 10.1016/j.otohns.2004.09.067. PMID 15577816

RESULTS

PARTICIPANT FLOW:
Groups:
- CT Scan (Sinus) Pre-tx: Sinus CT scan performed at initial otolaryngology (ear, nose, and throat)visit. This study was riskless, and was meant to study the timing of a test (CT) so there were no patients subjected to risk of an adverse event.
- CT Scan (Sinus) Post-tx: Sinus CT scan performed after 3-4 weeks of antibiotic treatment and any other indicated medical treatment(s), per insurance company guidelines. This study was riskless, and was meant to study the timing of a test (CT) so there were no patients subjected to risk of an adverse event.
Period: Overall Study
Arm/Group | CT Scan (Sinus) Pre-tx | CT Scan (Sinus) Post-tx
Started | 20 | 20
Completed | 20 | 14
Not Completed | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT Scan (Sinus) Pre-tx | CT Scan (Sinus) Post-tx | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (13.5) | 38.9 (11.6) | 39 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Compliance With Medical Recommendations
Description: Number of participants in each group who complied with medical advice given at the initial appointment.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | CT Scan (Sinus) Pre-tx | CT Scan (Sinus) Post-tx
Number analyzed (Participants) | 20 | 20
participants | 20 | 10

2. Primary Outcome: Number of Participants Having a CT Done
Description: Total number of participants having a CT scan (sinus) done in each of the two groups over the study interval.
Time Frame: 8 weeks
Population: Per protocol; this was a nonpowered convenience sample
Measure: Number; unit: participants
Arm/Group | CT Scan (Sinus) Pre-tx | CT Scan (Sinus) Post-tx
Number analyzed (Participants) | 20 | 20
participants | 20 | 9

ADVERSE EVENTS:
Arm/Group | CT Scan (Sinus) Pre-tx | CT Scan (Sinus) Post-tx
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes